CLINICAL TRIAL: NCT02585687
Title: Liver Perfusion MRI With Quantification of Tumoral Perfusion for Early Assessment of the Response of Antiangiogenics Treatments in Hepatocellular Carcinoma
Acronym: ETAFIRM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: problems with enrollment
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2011.693
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2015-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver Perfusion MRI, Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- liver Perfusion MRI (Experimental): liver perfusion MRI will be performed in patients to assess the early response (7 days) to antiangiogenic treatments
  Interventions: Device: liver Perfusion MRI

INTERVENTIONS:
Device: liver Perfusion MRI

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common cancer worldwide with an incidence of 500 000 cases per year. HCC most commonly appears in a context of liver chronic disease (patient with chronic viral hepatitis (hepatitis B or hepatitis C) or with cirrhosis). Surgical resection and liver transplantation concern patients with early stage and are the only curative treatments. Transcatheter arterial chemoembolization, Radiation Therapy and antiangiogenics treatments concern patients with inoperable lesions (palliative treatments).

Antiangiogenic treatments enable to inhibit the angiogenesis process and thus interrupt the blood supply to the tumor. In clinical practice, the efficacy of anti-angiogenic agents is usually assessed by methods based on morphological medical imaging. The measures of each target lesion are obtained by Response Evaluation Criteria In Solid Tumor (RECIST) criteria and WHO.

However, these morphological measures are not fully evaluated. An alternative to these is the functional medical imaging which assess changes before that a diminution of tumor size is detectable. Since these treatments induce generally necrosis without modification of initial tumor size, the new technologies of functional medical imaging are particularly adapted to an early evaluation of the response to treatments which may improve patient management.

In this context, liver Perfusion MRI needs to be assessed in its capacities to early predict the response of antiangiogenic treatments.

Positive results will enable to adapt therapy in order to improve overall survival of patients and avoid expensive treatments which may turn out to be inefficient and generating important side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocellular carcinoma diagnosis according to Barcelona Clinic Liver Cancer (BCLC) staging and European Association for Study of Liver (EASL) criteria or histologically confirmed diagnosis (biopsy).
* Patients with untreated hepatocellular carcinoma, not suitable for curative treatment and having an anti-angiogenic treatment.
* Patients with no contra-indication to sorafenib treatment
* The previous treatment with surgery, chemo-embolization, radiofrequency, or conformal radiotherapy are not contra-indications to the inclusion
* Patients agreeing to participate (signed inform consent)

Exclusion Criteria:

* Patients with contra-indication to sorafenib treatment
* MRI contra-indication: ferromagnetic material, pacemaker, intraocular foreign bodies, claustrophobia, creatinine clearance below 30 ml / min by Modification of Diet in Renal Disease (MDRD) method
* True allergy to gadobenate dimeglumine
* Patients suffering from acute renal failure or chronic severe (GFR <30 ml/min/1, 73 m²) and patients suffering from acute renal failure (regardless of severity) due to an hepatorenal syndrome
* Pregnancy or breast-feeding
* Refusal to sign the informed consent
* Patient has already been included in another study that could interfere with the results of the study. - Patients not affiliated to either the French social security system or an European health insurance.
* All persons deprived of liberty by a judicial or administrative law, patients hospitalized without consent under Articles L. 3212-1 and L. 3213-1 which are not covered by the provisions of Article L. 1121-8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Response to angiogenic treatment following morphological RECIST criteria | 7 days after angiogenic treatment
Survival without tumor progression | 7 days after angiogenic treatment
Global survival | 7 days after angiogenic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Agnès RODE, MD, PhD, Principal Investigator — Service d'Imagerie Médicale, Hôpital Croix-Rousse, Hospices Civils de Lyon
Locations (1):
- Service d'Imagerie, MédicaleHôpital Croix-Rousse, Lyon, France